CLINICAL TRIAL: NCT00604409
Title: Phase I Study of Capecitabine in Combination With SIR-Spheres in Patients With Advanced Cancer
Brief Title: Study of Capecitabine in Combination With SIR-Spheres in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCCC04043; NCI-2010-01936 (Registry Identifier: NCI Clinical Trials Reporting Office)
Record Dates: First submitted 2007-12-28; First posted 2008-01-30 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Metastatic Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Sirtuins; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (SIRT and capecitabine) (Experimental): Patients receive capecitabine PO twice daily on days 1-14. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients undergo SIRT on day 2 and may undergo a second course of SIRT on day 58.
  Interventions: Radiation: SIRT; Drug: capecitabine

INTERVENTIONS:
Radiation: SIRT — Undergo SIRT
  Other Names: selective internal radiation therapy
Drug: capecitabine — Given PO
  Other Names: CAPE, Ro 09-1978/000, Xeloda

SUMMARY:
This trial is testing the safety of combining the oral chemotherapy drug capecitabine with radio-labeled microspheres injected directly into the liver.

DETAILED DESCRIPTION:
Patients with adequate liver function and performance status in whom liver-directed therapy and capecitabine would be appropriate are eligible for this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adequate liver function
* Adequate performance status

Exclusion Criteria:

* Significant extrahepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-04; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety, toxicity, and recommended phase II dose (RPTD) of capecitabine when administered concurrently with SIR-Spheres in patients with advanced cancer. | ongoing

SECONDARY OUTCOMES:
Efficacy | response rate

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Cohen, M.D., Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States